CLINICAL TRIAL: NCT06795386
Title: Determining Mechanisms of Pain Reduction in Chronic Widespread Pain After Rapid Weight Loss in Non-Hispanic Black and Hispanic/Latino/a/x Adults
Brief Title: Chronic Widespread Pain After Rapid Weight Loss in Non-Hispanic Black and Hispanic/Latino/a/x Adults
Status: Recruiting | Type: Observational
Sponsor: New York University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Other Study IDs: i21-01652; 1K23AR080846-01A1 (NIH); 5K23AR080846-02 (NIH)
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Chronic Pain, Widespread; Obesity; Bariatric Surgery Candidate
Keywords: chronic pain, adult obesity, pain equity, rehabilitation
MeSH Terms: conditions — Chronic Pain; Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Racialized adults with chronic widespread pain: Adults who self-identify as non-Hispanic Black and/or Hispanic/Latino by the U.S. Census have elected to undergo bariatric surgery. All study participants will undergo bariatric surgery as part of the standard of care for surgical weight loss and will not be randomized to any other placebo or control interventions for weight loss or pain.
  Interventions: Procedure: Bariatric Surgery

INTERVENTIONS:
Procedure: Bariatric Surgery — Participants will include people with chronic widespread pain who will undergo bariatric surgery. All participants will receive this intervention and will not be randomized to this or other interventions.

SUMMARY:
The goal of this observational study is to learn if surgical weight loss can improve chronic widespread pain in people living with higher BMI who self-identify as Hispanic/Latino ethnicity or non-Hispanic Black based on the United States census racial categories. The main questions the study aims to answer are:

1. Do pain at rest (primary outcome) and movement-evoked pain (secondary outcome) improve after bariatric surgery?
2. Do pain processing and joint function change after bariatric surgery?
3. Are pain processing and joint function associated with clinically significant pain change after surgical weight loss?

Researchers will compare pain and function before and 6 months after bariatric surgery in a single cohort.

DETAILED DESCRIPTION:
The central hypothesis that will be tested is that pain at rest (primary outcome) and movement-evoked pain (MEP, secondary outcome) will decrease after bariatric surgery. We will also determine if pain reduction will be mediated by improved pain modulation and select joint motion and loading variables. The study will feature a prospective, observational quasi-experimental cohort study design for within-group analyses of pain at rest and MEP using the Numeric Pain Rating Scale (NPRS) and other exploratory outcomes before and 6 months after bariatric surgery. Pain at rest and MEP at 3 months after bariatric surgery are secondary endpoints. All participants will attend two in-person study visits and one off-site (remote) visit. Laboratory-based measurement and evaluation of pain and weight loss will be conducted during two in-person visits 1-3 months before bariatric surgery (Visit 1) at 6 months (Visit 3, primary endpoint). Pain surveys, weight measurements, and health questionnaires will be administered online or via telephone 3 months after surgery to assess acute post-surgical pain, weight loss, and other secondary and exploratory health outcomes (Visit 2). Descriptive analyses of all data will be performed by the NYU Biostatistics Resource directed by Dr. Huilin Li.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as Black/African American or Hispanic/Latino ethnicity based on the U.S Census racial categories
* Eligible candidates for bariatric surgery (BMI greater than or equal to 40 or BMI greater than or equal to 35 with comorbidity
* Meets criteria for chronic widespread pain (CWP) based on the following:

  1. self-reported pain at 3 or more anatomical sites
  2. painful regions on both sides of the body
  3. self-reported pain intensity at rest of 3 out of 10 or higher using the Numeric Pain Rating Scale (NPRS) or equivalent
* Conversational language fluency in English or Spanish
* Able to give voluntary, written informed consent to participate
* Able to walk independently or with a cane prior to study enrollment

Exclusion Criteria:

* Prospective participants with a previous history of bariatric surgery
* Have acute pain (pain for less than 6 weeks) at 1 month prior to study enrollment
* Have a systemic autoimmune disorder or immunodeficiency
* Have an unstable psychological condition
* Are non-ambulatory or ambulate with an assistive device other than a cane
* Pain localized to surgical sites at 3 months post-surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: New York City Health + Hospitals/Bellevue Hospital Center Bariatric Surgery Clinic
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Intensity at Rest as Assessed Using the Numeric Pain Rating Scale (NPRS) | At baseline, 3 months (secondary endpoint), and 6 months (primary endpoint) post-surgery
  Participant-reported pain intensity at rest will be assessed post-surgery using the Numeric Pain Rating Scale (NPRS). The NPRS is an ordinal scale with scores ranging from 0-10. Zero is indicative of no pain and 10 indicates the worst pain imaginable.

SECONDARY OUTCOMES:
Change in Movement-Evoked Pain Intensity as Assessed Using the Numeric Pain Rating Scale (NPRS) | Baseline, 6 months post-surgery
  Participant-reported pain during functional movement tasks will be assessed using the Numeric Pain Rating Scale (NPRS). The NPRS is an ordinal scale with scores ranging from 0-10. Zero is indicative of no pain and 10 indicates the worst pain imaginable.

OTHER OUTCOMES:
Mean Body Weight at Baseline | Baseline (pre-surgery)
  Body Weight will be measured in kilograms using a digital scale. Two measurements will be taken. A third measurement will be taken if these measurements differ by 0.5 kg or more. The average of the measurements will be included in all statistical analyses.
Mean Body Weight at 3 Months Post-surgery | 3 Months Post-surgery
  Participant-reported body weight measured in kilograms.
Mean Body Weight at 6 Months Post-surgery | 6 Months Post-surgery
  Body Weight will be measured in kilograms using a digital scale. Two measurements will be taken. A third measurement will be taken if these measurements differ by 0.5 kg or more. The average of the measurements will be included in all statistical analyses.
Height - Standing Height at Baseline | Baseline (pre-surgery)
  Standing height will be measured using a stadiometer from the crown of the participant's head to the lowest point on their heels. Two measurements of standing height will be taken in centimeters. A third measurement will be taken if these measurements differ by 1.0 or more. The average of the measurements will be used in all statistical analyses.
Waist Circumference at Baseline | Baseline (pre-surgery)
  Waist circumference is the measurement of the waist at the apex of the pelvis (ilium) in centimeters using a tape measure. Two measurements will be taken. A third measurement will be taken if there is a 1.0-centimeter or greater difference between the previous measurements. The average of the measurements will be used in all statistical analyses.
Waist Circumference at 6 Months Post-Surgery | 6 Months Post-surgery
  Waist circumference is the measurement of the waist at the apex of the pelvis (ilium) in centimeters using a tape measure. Two measurements will be taken. A third measurement will be taken if there is a 1.0-centimeter or greater difference between the previous measurements. The average of the measurements will be used in all statistical analyses.
Body Mass Index (BMI) at Baseline | Baseline (pre-surgery)
  Body Mass Index is the ratio of a person's body weight in kilograms divided by the squared value of their height in meters. BMI is used as a screening measure of individual and population health. BMI values greater than 30 indicate adult obesity.
Body Mass Index (BMI) at 3 Months Post-Surgery | 3 Months Post-surgery
  Body Mass Index is the ratio of a person's body weight in kilograms divided by the squared value of their height in meters. BMI is used as a screening measure of individual and population health. BMI values greater than 30 indicate adult obesity.
Body Mass Index (BMI) at 6 Months Post-surgery | 6 Months Post-surgery
  Body Mass Index is the ratio of a person's body weight in kilograms divided by the squared value of their height in meters. BMI is used as a screening measure of individual and population health. BMI values greater than 30 indicate adult obesity.
Percentage of Total Weight Loss (%TWL) at 3 Months Post-Surgery | 3 Months Post-surgery
  The percentage of total weight loss is the percentage of weight after bariatric surgery compared with pre-surgical weight. It is calculated as (baseline weight - current weight) / (baseline weight) × 100.
Percentage of Total Weight Loss (%TWL) at 6 Months Post-Surgery | 6 Months Post-surgery
  The percentage of total weight loss is the percentage of weight after bariatric surgery compared with pre-surgical weight. It is calculated as (baseline weight - current weight) / (baseline weight) × 100.
Knee Joint Range of Motion Using Goniometry at Baseline | Baseline (pre-surgery)
  Range of motion is the angle through which a joint moves. Knee flexion and extension will be measured bilaterally in degrees using a standard long arm goniometer. Two measurements of maximum knee flexion and knee extension angles will be taken. A third measurement will be taken if there is a difference of 5 degrees or more between the previous measurements. The average of the measurements will be included in all statistical analyses.
Knee Joint Range of Motion Using Goniometry at 6 Months Post-Surgery | 6 Months Post-surgery
  Range of motion is the angle through which a joint moves. Knee flexion and extension will be measured bilaterally in degrees using a standard long arm goniometer. Two measurements of maximum knee flexion and knee extension angles will be taken. A third measurement will be taken if there is a difference of 5 degrees or more between the previous measurements. The average of the measurements will be included in all statistical analyses.
Lumbar Spine Range of Motion at Baseline | Baseline (pre-surgery)
  Range of motion is the angle through which a joint moves. Lumbar spine flexion and extension will be measured in degrees using two (2) bubble inclinometers place at the cervical (neck) and lumbar (low back) spine. The data will be the calculated difference between the bubble inclinometer measurements at the two sites. Two measurements of maximum lumbar flexion and extension angles will be taken. A third measurement will be taken if the previous two differ by 5 degrees or more, and the average of the measurements will be included in all statistical analyses.
Lumbar Spine Range of Motion at 6 Months Post-surgery | 6 Months Post-surgery
  Range of motion is the angle through which a joint moves. Lumbar spine flexion and extension will be measured in degrees using two (2) bubble inclinometers place at the cervical (neck) and lumbar (low back) spine. The data will be the calculated difference between the bubble inclinometer measurements at the two sites. Two measurements of maximum lumbar flexion and extension angles will be taken. A third measurement will be taken if the previous two differ by 5 degrees or more, and the average of the measurements will be included in all statistical analyses.
Physical Function as Assessed Using the Six-Minute Walk Test (6MWT) at Baseline | Baseline (pre-surgery)
  The Six-Minute Walk Test (6MWT) is a standardized assessment of aerobic capacity, cardiovascular endurance, and physical function. This assessment measures the maximum distance a person can walk as quickly as possible in 6 minutes. The distance walked in meters will be included in all statistical analyses.
Physical Function as Assessed Using the Six-Minute Walk Test (6MWT) at 6 Months Post-surgery | 6 Months Post-surgery
  The Six-Minute Walk Test (6MWT) is a standardized assessment of aerobic capacity, cardiovascular endurance, and physical function. This assessment measures the maximum distance a person can walk as quickly as possible in 6 minutes. The distance walked in meters will be included in all statistical analyses.
Physical Function as Assessed Using the Five Time Sit-to-Stand Test (FTSTS) at 6 Months Post-Surgery | 6 Months Post-surgery
  This is a standardized clinical assessment of functional lower extremity strength. It is measured as the time (seconds) it takes for participants to complete the transition from sitting in a chair to a standing position as quickly as possible. The time in seconds will be included in all statistical analyses.
Physical Function as Assessed Using the Five Time Sit-to-Stand Test (FTSTS) at Baseline | Baseline (pre-surgery)
  The Five Time Sit-to-Stand Test (FTSTS) is a standardized clinical assessment of functional lower extremity strength. It is measured as the time (seconds) it takes for participants to complete the transition from sitting in a chair to a standing position as quickly as possible. The time in seconds will be included in all statistical analyses.
Pain Sensitivity as Assessed Using Pressure Pain Threshold at Baseline | Baseline (pre-surgery)
  Pressure pain threshold is a measure of static pain sensitivity. Pressure pain threshold will be measured 3 times using a pressure algometer at 3 anatomical locations: the upper trapezius, the medial side of the knee joint, and the lumbar spine. The force in kilopascals at which participants indicate a transition from a pressure sensation to pain greater than or equal to 1 out of 10 will be recorded. The mean force values for all trials and anatomical sites will be used in a statistical analyses.
Pain Sensitivity as Assessed Using Pressure Pain Threshold at 6M Post-surgery | 6 Months Post-surgery
  Pressure pain threshold is a measure of static pain sensitivity. Pressure pain threshold will be measured 3 times using a pressure algometer at 3 anatomical locations: the upper trapezius, the medial side of the knee joint, and the lumbar spine. The force in kilopascals at which participants indicate a transition from a pressure sensation to pain greater than or equal to 1 out of 10 will be recorded. The mean force values for all trials and anatomical sites will be used in a statistical analyses.
Pain Sensitivity as Assessed Using Conditioned Pain Modulation at Baseline | Baseline (pre-surgery)
  Conditioned pain modulation is a measure of dynamic pain sensitivity in which the application of second noxious stimulus (conditioning stimulus) reduces pain intensity ratings from an initial noxious stimulus (test stimulus). The test stimulus in the current study paradigm will be a standardized and calibrated mechanical stimulus and the conditioning stimulus will be thermal (cold water immersion). Pain intensity ratings and mechanical force in kilopascals will be recorded, and mean values will be used in all statistical analyses.
Pain Sensitivity as Assessed Using Conditioned Pain Modulation at 6M Post-surgery | 6 Months Post-surgery
  Conditioned pain modulation is a measure of dynamic pain sensitivity in which the application of second noxious stimulus (conditioning stimulus) reduces pain intensity ratings from an initial noxious stimulus (test stimulus). The test stimulus in the current study paradigm will be a standardized and calibrated mechanical stimulus and the conditioning stimulus will be thermal (cold water immersion). Pain intensity ratings and mechanical force in kilopascals will be recorded, and mean values will be used in all statistical analyses.
Pain Sensitivity as Assessed Using Temporal Summation at 6M Post-surgery | 6 Months Post-surgery
  Conditioned pain modulation is a measure of dynamic pain sensitivity in which the pain increases after the application of repetitive, noxious stimuli. The stimulus in the current study paradigm will be the application of a standardized and calibrated probe (128 nM) as the mechanical stimulus. The probe will be applied to 3 anatomical sitePain intensity ratings before and after the 10th applicatio will be recorded, and mean values will be used in all statistical analyses.
Pain Sensitivity as Assessed Using Temporal Summation at Baseline | Baseline
  Conditioned pain modulation is a measure of dynamic pain sensitivity in which the pain increases after the application of repetitive, noxious stimuli. The stimulus in the current study paradigm will be the application of a standardized and calibrated probe (128 nM) as the mechanical stimulus. The probe will be applied to 3 anatomical sitePain intensity ratings before and after the 10th applicatio will be recorded, and mean values will be used in all statistical analyses.
Pain Intensity and Interference as Assessed Using the Brief Pain Inventory Short Form (BPI-SF) at Baseline | Baseline (pre-surgery)
  The Brief Pain Inventory Short Form (BPI-SF) is a 9-item self-assessment with 2 subscales that measure pain intensity and how pain interferes with daily activities. The BPI-SF Pain Severity subscale ranges from 0 ("no pain") to 10 ("Pain As Bad As You Can Imagine"). The Pain Severity subscale score is the mean of 4 items. The Pain Interference subscale score is the mean of 7 items. The BPI-SF will be administered electronically or using written forms in either English or Spanish.
Pain Intensity and Interference as Assessed Using the Brief Pain Inventory Short Form (BPI-SF) at 3 Months Post-surgery | 3 Months Post-surgery
  The Brief Pain Inventory Short Form (BPI-SF) is a 9-item self-assessment with 2 subscales that measure pain intensity and how pain interferes with daily activities. The BPI-SF Pain Severity subscale ranges from 0 ("no pain") to 10 ("Pain As Bad As You Can Imagine"). The Pain Severity subscale score is the mean of 4 items. The Pain Interference subscale score is the mean of 7 items. The BPI-SF will be administered electronically or using written forms in either English or Spanish.
Pain Intensity and Interference as Assessed Using the Brief Pain Inventory Short Form (BPI-SF) at 6 Months Post-surgery | 6 Months Post-surgery
  The Brief Pain Inventory Short Form (BPI-SF) is a 9-item self-assessment with 2 subscales that measure pain intensity and how pain interferes with daily activities. The BPI-SF Pain Severity subscale ranges from 0 ("no pain") to 10 ("Pain As Bad As You Can Imagine"). The Pain Severity subscale score is the mean of 4 items. The Pain Interference subscale score is the mean of 7 items. The BPI-SF will be administered electronically or using written forms in either English or Spanish.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - NYU Steinhardt Arthur J. Nelson Laboratory, New York, New York
  - New York City Health + Hospitals/Bellevue Hospital, New York, New York
  - NYU CTSI Clinical Research Center, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided
Since we are working with a document-diverse population, we will consult with university and local officials to determine the most appropriate course of action.